CLINICAL TRIAL: NCT02723630
Title: A Randomized, Three-treatment, Three-period, Six-sequence Crossover, Single-center, Bioequivalence Study to Evaluate the Impact of Varying Crystalline Polymorph Forms for the Commercial Oral Capsule Formulation of 10-mg Lenvatinib in Healthy Volunteers
Brief Title: Bioequivalence Study to Evaluate the Impact of Varying Crystalline Polymorph Forms for the Commercial Oral Capsule Formulation of 10-mg Lenvatinib in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E7080-A001-008
Record Dates: First submitted 2015-10-15; First posted 2016-03-30 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2018-03

CONDITIONS: Healthy Volunteers
Keywords: Bioequivalence; Lenvatinib; Healthy Volunteers; Lenvima; E7080
MeSH Terms: interventions — lenvatinib

ARMS (6):
- Sequence A: (Experimental): Participants will receive one dose of Treatment 1 followed by one dose of Treatment 2, then one dose of Treatment 3
  Interventions: Drug: Lenvatinib 10 mg
- Sequence B (Experimental): Participants will receive one dose of Treatment 2, followed by one dose of Treatment 3, then one dose of Treatment 1
  Interventions: Drug: Lenvatinib 10 mg
- Sequence C (Experimental): Participants will receive one dose of Treatment 3, followed by one dose of Treatment 1, then one dose of Treatment 2
  Interventions: Drug: Lenvatinib 10 mg
- Sequence D (Experimental): Participants will receive one dose of Treatment 3, followed by one dose of Treatment 2, then one dose of Treatment 1
  Interventions: Drug: Lenvatinib 10 mg
- Sequence E (Experimental): Participants will receive one dose of Treatment 1, followed by one dose of Treatment 3, then one dose of Treatment 2
  Interventions: Drug: Lenvatinib 10 mg
- Sequence F (Experimental): Participants will receive one dose of Treatment 2, followed by one dose of Treatment 1, then one dose of Treatment 3
  Interventions: Drug: Lenvatinib 10 mg

INTERVENTIONS:
Drug: Lenvatinib 10 mg — Treatment 1: low Type-C crystal level <12%
  Treatment 2: reference* Type-C crystal level 12% to 26%
  Treatment 3: high Type-C crystal level >26%
  Other Names: E7080;Lenvima

SUMMARY:
This will be a randomized, single dose, open-label, three-treatment period crossover study in healthy participants to determine whether 2 test lots of 10-mg capsules that vary by the level of lenvatinib Type-C crystal are bioequivalent to a reference lot of 10-mg capsules.

DETAILED DESCRIPTION:
The study will consist of 2 phases: Prerandomization and Randomization. The Prerandomization Phase will have 2 periods: Screening and Baseline. The Randomization Phase will consist of three 6-day long Treatment Periods with each Treatment Period separated by a 1-day long Baseline. Sixty participants will be evenly randomized to 1 of 6 possible treatment sequences (A, B, C, D, E, or F). The 3 treatments vary by the level of crystalline polymorph Type-C present in the drug product batch used in each arm, respectively: Treatment 1 - low Type-C crystal level less than 12%; Treatment 2 - reference Type-C crystal level 12% to 26%; and Treatment 3 - high Type-C crystal level greater than 26%.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female participants age greater than or equal to 18 years and less than or equal to 55 years old
2. Nonsmokers or smokers who smoke no more than 10 cigarettes per day
3. BMI greater than or equal to 18 and less than or equal to 32 kg/m2 at Screening
4. Females must not be lactating or pregnant at Screening or Baseline (as documented by a negative beta-human chorionic gonadotropin)
5. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing)
6. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days before study entry and must agree to use a highly effective method of contraception (e.g., total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 30 days after study drug discontinuation. If currently abstinent, the participant must agree to use a double-barrier method as described above if she becomes sexually active during the study period or for 30 days after study drug discontinuation. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation.
7. Male participants must have had a successful vasectomy (confirmed azoospermia) or they and their female partners must meet the criteria above (i.e., not of childbearing potential or practicing highly effective contraception throughout the study period and for 30 days after study drug discontinuation). No sperm donation is allowed during the study period and for 30 days after study drug discontinuation.
8. Provide written informed consent

Exclusion Criteria:

1. Clinically significant illness that requires medical treatment within 8 weeks of Screening or a clinically significant infection that requires medical treatment within 4 weeks of dosing
2. Evidence of disease that may influence the outcome of the study within 4 weeks prior to dosing, e.g., psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism
3. Any history of GI surgery that may affect pharmacokinetic profiles of lenvatinib e.g., hepatectomy, nephrotomy, digestive organ resection known at Screening or Baseline
4. Any clinically abnormal symptom or organ impairment found by medical history, physical examinations, vital signs, ECG findings, or laboratory test results that require medical treatment at Screening or Baseline
5. Blood pressure measurements of greater than 150/90 mm Hg. Confirmation should be obtained by performing three measurements (at least 5 minutes apart) to yield a mean value. Participants may be enrolled if they are on a stable dose of a single antihypertensive drug at least 30 days prior to the first dose of study drug and do not intend to change the dose or drug during the study.
6. A prolonged QTcF interval (QTcF greater than 450 ms) demonstrated on ECG at Screening or Baseline
7. Known history of clinically significant drug allergy at Screening or Baseline
8. Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening or Baseline or with a known history of sensitivity to any of the components of the test products
9. Known to be human immunodeficiency virus positive at Screening
10. Active viral hepatitis (A, B, or C) as demonstrated by positive serology at Screening
11. History of drug or alcohol dependency or abuse within the 2 years prior to Screening or a positive urine drug test at Screening or Baseline
12. Intake of grapefruit or grapefruit-containing beverages or food within 72 hours prior to dosing
13. Intake of medications known to be strong inhibitors or inducers of CYP450 3A4 metabolizing enzymes within 2 weeks prior to dosing
14. Currently enrolled in another clinical trial or used any investigational drug or device within 30 days preceding informed consent
15. Receipt of blood products within 4 weeks, or donation of blood within 8 weeks, or donation of plasma within 1 week of dosing
16. Engagement in strenuous exercise within 2 weeks prior to check-in (e.g., marathon runners, weight lifters)
17. Any condition that would make the participant, in the opinion of the investigator or sponsor unsuitable for the study or not likely to complete the study for any reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence A: The Randomization Phase consisted of three 6-day long Treatment Periods with each Period separated by a 1-day long Baseline. Sixty participants were evenly randomized to one of 6 possible treatment sequences (A, B, C, D, E, or F). Participants in Sequence A were administered lenvatinib with 240 mL of water in the following sequence; Treatment 1 (low Crystal form Type-C level <4%), Treatment 2 (reference* Crystal form Type-C level 15%, *reference range determined from clinical batches), and Treatment 3 (high Crystal form Type-C level 38%) on the morning of Days 1, 8, and 15 following an overnight fast of at least 10 hours. No food was allowed for at least 4 hours postdose. Water was allowed ad libitum except for the period beginning 1 hour before and lasting until 1 hour after treatment. Treatments were administered at the same time on the 3 mornings. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Sequence B: The Randomization Phase consisted of three 6-day long Treatment Periods with each Period separated by a 1-day long Baseline. Sixty participants were evenly randomized to one of 6 possible treatment sequences (A, B, C, D, E, or F). Participants in Sequence B were administered lenvatinib with 240 mL of water in the following sequence; Treatment 2 (reference* Crystal form Type-C level 15%, *reference range determined from clinical batches), Treatment 3 (high Crystal form Type-C level 38%), and Treatment 1 (low Crystal form Type-C level <4%), on the morning of Days 1, 8, and 15 following an overnight fast of at least 10 hours. No food was allowed for at least 4 hours postdose. Water was allowed ad libitum except for the period beginning 1 hour before and lasting until 1 hour after treatment. Treatments were administered at the same time on the 3 mornings. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Sequence C: The Randomization Phase consisted of three 6-day long Treatment Periods with each Period separated by a 1-day long Baseline. Sixty participants were evenly randomized to one of 6 possible treatment sequences (A, B, C, D, E, or F). Participants in Sequence C were administered lenvatinib with 240 mL of water in the following sequence; Treatment 3 (high Crystal form Type-C level 38%), Treatment 1 (low Crystal form Type-C level <4%), and Treatment 2 (reference* Crystal form Type-C level 15%, *reference range determined from clinical batches), on the morning of Days 1, 8, and 15 following an overnight fast of at least 10 hours. No food was allowed for at least 4 hours postdose. Water was allowed ad libitum except for the period beginning 1 hour before and lasting until 1 hour after treatment. Treatments were administered at the same time on the 3 mornings. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Sequence D: The Randomization Phase consisted of three 6-day long Treatment Periods with each Period separated by a 1-day long Baseline. Sixty participants were evenly randomized to one of 6 possible treatment sequences (A, B, C, D, E, or F). Participants in Sequence D were administered lenvatinib with 240 mL of water in the following sequence; Treatment 3 (high Crystal form Type-C level 38%), Treatment 2 (reference* Crystal form Type-C level 15%, *reference range determined from clinical batches), and Treatment 1 (low Crystal form Type-C level <4%), on the morning of Days 1, 8, and 15 following an overnight fast of at least 10 hours. No food was allowed for at least 4 hours postdose. Water was allowed ad libitum except for the period beginning 1 hour before and lasting until 1 hour after treatment. Treatments were administered at the same time on the 3 mornings. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Sequence E: The Randomization Phase consisted of three 6-day long Treatment Periods with each Period separated by a 1-day long Baseline. Sixty participants were evenly randomized to one of 6 possible treatment sequences (A, B, C, D, E, or F). Participants in Sequence E were administered lenvatinib with 240 mL of water in the following sequence; Treatment 1 (low Crystal form Type-C level <4%), Treatment 3 (high Crystal form Type-C level 38%), and Treatment 2 (reference* Crystal form Type-C level 15%, *reference range determined from clinical batches), on the morning of Days 1, 8, and 15 following an overnight fast of at least 10 hours. No food was allowed for at least 4 hours postdose. Water was allowed ad libitum except for the period beginning 1 hour before and lasting until 1 hour after treatment. Treatments were administered at the same time on the 3 mornings. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
- Sequence F: The Randomization Phase consisted of three 6-day long Treatment Periods with each Period separated by a 1-day long Baseline. Sixty participants were evenly randomized to one of 6 possible treatment sequences (A, B, C, D, E, or F). Participants in Sequence F were administered lenvatinib with 240 mL of water in the following sequence; Treatment 2 (reference* Crystal form Type-C level 15%, *reference range determined from clinical batches), Treatment 1 (low Crystal form Type-C level <4%), and Treatment 3 (high Crystal form Type-C level 38%), on the morning of Days 1, 8, and 15 following an overnight fast of at least 10 hours. No food was allowed for at least 4 hours postdose. Water was allowed ad libitum except for the period beginning 1 hour before and lasting until 1 hour after treatment. Treatments were administered at the same time on the 3 mornings. On dosing days, all participants observed identical schedules with respect to fasting before dosing and timing of postdose meals.
Period: Intervention Period 1
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Sequence E | Sequence F
Started | 10 | 10 | 10 | 10 | 10 | 10
Completed | 9 | 10 | 10 | 10 | 10 | 10
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Period: Intervention Period 2
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Sequence E | Sequence F
Started | 9 | 10 | 10 | 10 | 10 | 10
Completed | 9 | 10 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention Period 3
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Sequence E | Sequence F
Started | 9 | 10 | 10 | 10 | 10 | 10
Completed | 9 | 9 | 10 | 10 | 10 | 10
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — consumption of restricted item | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) included all participants who received at least one dose of study drug and had at least one postdose safety assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Sequence E | Sequence F | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.1 (9.55) | 45.1 (10.72) | 36.3 (13.41) | 40.4 (10.80) | 31.7 (10.36) | 37.8 (12.06) | 39.4 (11.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 2 | 2 | 2 | 15
  Male | 6 | 7 | 8 | 8 | 8 | 8 | 45

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Zero Time (Predose) to Time of Last Quantifiable Concentration (AUC(0-t))
Description: Blood samples (6 mL each) were collected at the following time points for each Period: 0 (Predose), 1, 2, 3, 4, 8, 12, 24, 48, 72, 96, and 120 hours postdose. The window for 0 to 12 hours was +/-2 minutes, for 24 hours was +/-5 minutes and for >24 hours was equal to +/-15 to 60 minutes. Plasma concentrations of lenvatinib were quantified by chromatography-mass spectrometry/mass spectrometry (LC-MS/MS) methodology using a previously validated assay. The lower limit of quantitation (LLOQ) for the assay was 0.25 ng/mL. AUC(0-t) was calculated by the linear-up log-down trapezoidal method. No concentration estimates were provided for missing sample values. Any sample with a missing value was treated as if the sample had not been scheduled for collection.
Time Frame: Periods 1, 2, and 3; 0 (Predose), 1, 2, 3, 4, 8, 12, 24, 48, 72, 96, and 120 hours postdose
Population: Pharmacokinetic (PK) analysis set included participants who had sufficient PK data to derive at least one PK parameter. Participants with a predose concentration >5% Cmax and participants who experienced emesis at or before two times median tmax were excluded from the data analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·hr/mL
Groups:
- Treatment 1: Low Crystal Form: Treatment 1: low Crystal form Type-C level < 4%
- Treatment 2: Reference Crystal Form: Treatment 2: reference (reference range determined from clinical batches) Crystal form Type-C level 15%
- Treatment 3: High Crystal Form: Treatment 3: high Crystal form Type-C level 38%
Arm/Group | Treatment 1: Low Crystal Form | Treatment 2: Reference Crystal Form | Treatment 3: High Crystal Form
Number analyzed (Participants) | 59 | 59 | 59
ng·hr/mL | 1010 (40.4) | 1010 (36.9) | 965 (39.3)
Statistical Analysis 1: Comparison: Treatment 1: Low Crystal Form vs Treatment 2: Reference Crystal Form; The effect of crystalline polymorph forms in the drug product on the PK parameters of lenvatinib was estimated using a mixed linear model of logarithmically transformed values of the primary PK parameters with fixed effects for treatment, period, and sequence and a random effect for participant within sequence; Test type: Superiority or Other; p = 0.8826, Mixed Models Analysis — P-value for the formulation; Geometric Least Square Mean Ratio = 100.52, 90% CI 2-sided [94.84 to 106.53] — Geometric LS Mean ratio was back-transformed least squares mean and mean treatment difference
Statistical Analysis 2: Comparison: Treatment 2: Reference Crystal Form vs Treatment 3: High Crystal Form; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1095, Mixed Models Analysis — P-value for formulation; Geometric Least Squares Mean Ratio = 96.03, 90% CI 2-sided [92.11 to 100.12] — Geometric LS Mean ratio was back-transformed least squares mean and mean treatment difference

2. Primary Outcome: Area Under the Concentration-Time Curve From Zero Time (Predose) Extrapolated to Infinite Time (AUC(0-inf))
Description: Blood samples (6 mL each) were collected at the following time points for each Period: 0 (Predose), 1, 2, 3, 4, 8, 12, 24, 48, 72, 96, and 120 hours postdose. The window for 0 to 12 hours was +/-2 minutes, for 24 hours was +/-5 minutes and for >24 hours was equal to +/-15 to 60 minutes. Plasma concentrations of lenvatinib were quantified by LC-MS/MS methodology using a previously validated assay. The LLOQ for the assay was 0.25 ng/mL. AUC(0-t) was calculated by the linear-up log-down trapezoidal method. AUC(0-inf) was calculate as follows; (AUC(0-inf)) = (AUC(0-t)) + (Ct/Kel), where Ct is the last measurable drug concentration and Kel is the elimination rate constant. The apparent first-order Kel was estimated, when possible, from the slope of the regression line for the terminal ln-linear concentration-time values.
Time Frame: Periods 1, 2, and 3; 0 (Predose), 2, 4, 8, 12, 24, 48, 72, 96, and 120 hours postdose.
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·hr/mL
Groups:
- Treatment 1: Low Crystal Form: Treatment 1: low Crystal form Type-C level <4%
- Treatment 2: Reference Crystal Form: Treatment 2: reference* Crystal form Type-C level 15%, *reference range determined from clinical batches
Arm/Group | Treatment 1: Low Crystal Form | Treatment 2: Reference Crystal Form | Treatment 3: High Crystal Form
Number analyzed (Participants) | 57 | 57 | 57
ng·hr/mL | 1030 (40.0) | 1020 (36.9) | 991 (39.0)
Statistical Analysis 1: Comparison: Treatment 1: Low Crystal Form vs Treatment 2: Reference Crystal Form; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8121, Mixed Models Analysis — P value for formulation; Geometric Least Squares Mean Ratio = 100.80, 90% CI 2-sided [95.31 to 106.61] — Geometric LS Mean ratio was back-transformed least squares mean and treatment difference mean
Statistical Analysis 2: Comparison: Treatment 2: Reference Crystal Form vs Treatment 3: High Crystal Form; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1630, Mixed Models Analysis — P value for formulation; Geometric Least Squares Mean Ratio = 96.51, 90% CI 2-sided [92.53 to 100.65] — Geometric LS Mean ratio was back-transformed least squares mean and treatment difference mean

3. Primary Outcome: Area Under the Concentration-Time Curve From Zero Time (Predose) to 24 Hours (AUC(0-24))
Description: Blood samples (6 mL each) were collected at the following time points for each Period: 0 (Predose), 1, 2, 3, 4, 8, 12, 24, 48, 72, 96, and 120 hours postdose. The window for 0 to 12 hours was +/-2 minutes, for 24 hours was +/-5 minutes and for >24 hours was equal to +/-15 to 60 minutes. Plasma concentrations of lenvatinib were quantified by LC-MS/MS methodology using a previously validated assay. The LLOQ for the assay was 0.25 ng/mL.
Time Frame: Periods 1, 2, and 3; 0 (Predose), 1, 2, 3, 4, 8, 12, and 24 hours postdose
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·hr/mL
Groups:
- Treatment 1: Low Crystal Form: Treatment 1: (low Crystal form Type-C level <4%)
- Treatment 2: Reference Crystal Form: Treatment 2: (reference* Crystal form Type-C level 15%, *reference range determined from clinical batches)
- Treatment 3: High Crystal Form: Treatment 3: (high Crystal form Type-C level 38%)
Arm/Group | Treatment 1: Low Crystal Form | Treatment 2: Reference Crystal Form | Treatment 3: High Crystal Form
Number analyzed (Participants) | 59 | 59 | 59
ng·hr/mL | 791 (47.4) | 792 (39.2) | 740 (43.5)
Statistical Analysis 1: Comparison: Treatment 1: Low Crystal Form vs Treatment 2: Reference Crystal Form; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9427, Mixed Models Analysis — P value for formulation; Geometric Least Squares Mean Ratio = 99.68, 90% CI 2-sided [92.45 to 107.47] — Geometric LS Mean ratio was back-transformed least squares mean and treatment difference mean
Statistical Analysis 2: Comparison: Treatment 2: Reference Crystal Form vs Treatment 3: High Crystal Form; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0403, Mixed Models Analysis — P value for formulation; Geometric Least Squares Mean Ratio = 93.50, 90% CI 2-sided [88.63 to 98.64] — Geometric LS Mean ratio was back-transformed least squares mean and treatment difference mean

4. Secondary Outcome: Area Under the Concentration-Time Curve From Zero Time (Predose) to 72 Hours (AUC(0-72))
Description: as for outcome 3
Time Frame: Periods 1, 2, and 3; 0 (Predose), 1, 2, 3, 4, 8, 12, 24, 48, and 72 hours postdose
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·hr/mL
Arm/Group | Treatment 1: Low Crystal Form | Treatment 2: Reference Crystal Form | Treatment 3: High Crystal Form
Number analyzed (Participants) | 59 | 59 | 59
ng·hr/mL | 975 (40.5) | 971 (36.7) | 923 (39.4)
Statistical Analysis 1: Comparison: Treatment 1: Low Crystal Form vs Treatment 2: Reference Crystal Form; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9373, Mixed Models Analysis — P value for formulation; Geometric Least Squares Mean Ratio = 100.29, 90% CI 2-sided [94.37 to 106.58] — Geometric LS Mean ratio was back-transformed least squares mean and treatment difference mean
Statistical Analysis 2: Comparison: Treatment 2: Reference Crystal Form vs Treatment 3: High Crystal Form; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0682, Mixed Models Analysis — P value for formulation; Geometric Least Squares Mean Ratio = 95.17, 90% CI 2-sided [91.03 to 99.50] — Geometric LS Mean ratio was back-transformed least squares mean and treatment difference mean

5. Secondary Outcome: Maximum Observed Concentration (Cmax) of Lenvatinib in Plasma
Description: as for outcome 3
Time Frame: Periods 1, 2, and 3; 0 (Predose), 1, 2, 3, 4, 8, 12, 24, 48, 72, 96, and 120 hours postdose
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment 1: Low Crystal Form | Treatment 2: Reference Crystal Form | Treatment 3: High Crystal Form
Number analyzed (Participants) | 59 | 59 | 59
ng/mL | 96.0 (64.0) | 97.1 (49.2) | 88.0 (57.7)
Statistical Analysis 1: Comparison: Treatment 1: Low Crystal Form vs Treatment 2: Reference Crystal Form; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8448, Mixed Models Analysis — P value for formulation; Geometric Least Squares Mean Ratio = 98.73, 90% CI 2-sided [88.57 to 110.06] — Geometric Least Squares Mean Ratio was back-transformed least squares mean and treatment difference mean
Statistical Analysis 2: Comparison: Treatment 2: Reference Crystal Form vs Treatment 3: High Crystal Form; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0498, Mixed Models Analysis — P value for formulation; Geometric Least Squares Mean Ratio = 90.64, 90% CI 2-sided [83.51 to 98.38] — Geometric LS Mean ratio was back-transformed least squares mean and treatment difference mean

6. Secondary Outcome: Time to Cmax (Tmax) for Lenvatinib
Description: as for outcome 3
Time Frame: Periods 1, 2, and 3; 0 (Predose), 1, 2, 3, 4, 8, 12, 24, 48, 72, 96, and 120 hours postdose
Population: PK analysis set
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment 1: Low Crystal Form | Treatment 2: Reference Crystal Form | Treatment 3: High Crystal Form
Number analyzed (Participants) | 59 | 59 | 59
Hours | 3.000 [1.00 to 12.00] | 3.000 [1.00 to 12.02] | 3.000 [2.00 to 12.02]

7. Secondary Outcome: Terminal Elimination Phase Half-life (t1/2)
Description: as for outcome 3
Time Frame: Periods 1, 2, and 3; 0 (Predose), 1, 2, 3, 4, 8, 12, 24, 48, 72, 96, and 120 hours postdose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Treatment 1: Low Crystal Form | Treatment 2: Reference Crystal Form | Treatment 3: High Crystal Form
Number analyzed (Participants) | 59 | 59 | 57
Hours | 24.1 (6.88) | 24.2 (6.23) | 23.5 (6.61)

8. Secondary Outcome: Number of Participants With Non-Serious Treatment-Emergent Adverse Events (TEAEs) and Serious Treatment-Emergent Adverse Events as a Measure of Safety and Tolerability of Lenvatinib
Description: Safety assessments consisted of monitoring and recording all adverse events (AEs) (serious and non-serious); regular monitoring of hematology, blood chemistry and urine values; periodic measurement of vital signs and electrocardiograms, performance of physical examinations. A TEAE was defined as an AE that emerges during treatment, having been absent at pretreatment (Baseline), or reemerges during treatment, having been present at pretreatment but stopped before treatment, or worsens in severity during treatment relative to the pretreatment state, when the AE is continuous. TEAEs considered by the investigator to be possibly or probably related to study drug, or TEAEs with missing causality, were included.
Time Frame: From date of first dose up to 30 days after the last dose of study treatment, up to approximately 2 months
Population: Safety analysis set (SAS) included the group of participants who received at least one dose of study drug and had at least one postdose safety assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment 1: Low Crystal Form | Treatment 2: Reference Crystal Form | Treatment 3: High Crystal Form
Number analyzed (Participants) | 59 | 59 | 59
Percentage of participants
  TEAEs | 23.7 | 23.7 | 20.3
  Treatment-related TEAEs | 18.6 | 15.2 | 16.9
  Severe TEAEs | 1.69 | 0 | 0
  Serious TEAEs | 1.69 | 0 | 0

ADVERSE EVENTS:
Time Frame: From date of first dose up to 30 days after the last dose of study treatment, up to approximately 2 months
Description: Treatment-emergent adverse events (TEAEs) were reported. TEAEs were defined as an adverse event (AE) that emerges during treatment, having been absent at pretreatment (Baseline), or reemerges during treatment, having been present at pretreatment but stopped before treatment, or worsens in severity during treatment relative to the pretreatment state, when the AE is continuous. AEs were graded on a 3-point scale (mild, moderate, severe). All serious AEs were reported.
Arm/Group | Treatment 1: Low Crystal Form | Treatment 2: Reference Crystal Form | Treatment 3: High Crystal Form
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 1/59 | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 14/59 | 14/59 | 12/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment 1: Low Crystal Form (N=59) | Treatment 2: Reference Crystal Form (N=59) | Treatment 3: High Crystal Form (N=59)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1: Low Crystal Form (N=59) | Treatment 2: Reference Crystal Form (N=59) | Treatment 3: High Crystal Form (N=59)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 1 | 0
Blood phosphorus increased (Investigations) | 1 | 0 | 0
Blood pressure increased (Investigations) | 2 | 2 | 1
Blood triglycerides increased (Investigations) | 0 | 1 | 0
Haematocrit decreased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 4 | 6
Lethargy (Nervous system disorders) | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Hypervigilance (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other